CLINICAL TRIAL: NCT01156805
Title: Assessment of an School-based Intervention in Eating Habits and Physical Activity in Schoolchildren: the AVall Study.
Acronym: AVALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AVALL
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2017-08

CONDITIONS: Obesity; Food Habits; Physical Activity
Keywords: Children; School-based program; Obesity
MeSH Terms: conditions — Obesity; Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational intervention, Control (Experimental): Experimental, intervention group has received specific educational training to improve food habits and physical activity during the period of the study.
  Interventions: Other: Educational program
- Educational program (No Intervention): No intervention has been made.

INTERVENTIONS:
Other: Educational program — The intervention consisted of the promotion of healthy eating habits and physical activity by means of the educational methodology Investigation, Vision, Action and Change (IVAC). At the beginning and at the end of 1st phase of the study (2006 and 2008) the weight and height of each child was measured in situ, while the families were given a self-report physical activity questionnaire and the Krece Plus quick test
  Arms: Educational intervention, Control

SUMMARY:
The objective of the study is to evaluate the efficacy of an intervention on food habits and physical activity in school-age children.

DETAILED DESCRIPTION:
A two-year cluster-randomised prospective study with two parallel arms was used to evaluate an intervention programme in children in their first year of primary schooling (5-6 years of age) in schools in the city of Granollers. The intervention consisted of the promotion of healthy eating habits and physical activity by means of the educational methodology Investigation, Vision, Action and Change (IVAC). At the beginning and at the end of the study (2006 and 2008) the weight and height of each child was measured in situ, while the families were given a self-report physical activity questionnaire and the Krece Plus quick test.

ELIGIBILITY:
Inclusion Criteria:

* Children born in 2000 who attended schools in Granollers City

Exclusion Criteria:

* Schoolchildren who need special diet for metabolic or digestive disorder, physical activity incapacity, no family acceptance or attendance to school was discontinued

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 509 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Assumpta Recasens, MD, Study Director — Hospital de Granollers

REFERENCES:
- [Derived] Recasens MA, Xicola-Coromina E, Manresa JM, Ullmo PA, Jensen BB, Franco R, Suarez A, Nadal A, Vila M, Recasens I, Perez MJ, Castell C, Llargues E. Impact of school-based nutrition and physical activity intervention on body mass index eight years after cessation of randomized controlled trial (AVall study). Clin Nutr. 2019 Dec;38(6):2592-2598. doi: 10.1016/j.clnu.2018.12.029. Epub 2019 Jan 24. PMID 30737048
- [Derived] Llargues E, Recasens MA, Manresa JM, Jensen BB, Franco R, Nadal A, Vila M, Recasens I, Perez MJ, Castell C. Four-year outcomes of an educational intervention in healthy habits in schoolchildren: the Avall 3 Trial. Eur J Public Health. 2017 Feb 1;27(1):42-47. doi: 10.1093/eurpub/ckw199. No abstract available. PMID 28177448

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In 2006, the 16 schools in Granollers were randomly distributed to the intervention or control group stratified according to public or semi-private status, number of first-year's classrooms and socioeconomic status of the local neighborhood.
Groups:
- Educational Intervention, Control: Experimental, intervention group has received educational training to improve food habits and physical activity
  Educational program: The intervention consisted of the promotion of healthy eating habits and physical activity by means of the educational methodology Investigation, Vision, Action and Change (IVAC). At the beginning and at the end of 1st phase of the study (2006 and 2008) the weight and height of each child was measured in situ, while the families were given a self-report physical activity questionnaire and the Krece Plus quick test
- Non Intervention: No intervention has been made.
Period: Overall Study
Arm/Group | Educational Intervention, Control | Non Intervention
Started | 237 | 272
Completed | 181 | 216
Not Completed | 56 | 56

BASELINE CHARACTERISTICS:
Groups:
- Educational Intervention, Control: Experimental, intervention group has received educational training to improve food habits and physical activity
  Educational program: The intervention consisted of the promotion of healthy eating habits and physical activity by means of the educational methodology Investigation, Vision, Action and Change (IVAC). At the beginning and at the end of 1st phase of the study (2006 and 2008) the weight and height of each child was measured in situ
- Total: Total of all reporting groups
Arm/Group | Educational Intervention, Control | Non Intervention | Total
Number analyzed (Participants) | 237 | 272 | 509
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 6.03 (0.3) | 6.03 (0.3) | 6.03 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 126 | 234
  Male | 129 | 146 | 275

OUTCOME MEASURES:

1. Primary Outcome: Anthropometric Variables
Description: BMI progression in the intervention and the control group. Secondary outcomes measured in this study were changes in eating habits and in physical activity.
Time Frame: every two years
Population: Qualitative variables are described in absolute and relative frequencies (percentages). Continuous variables are described as mean and SD.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Educational Intervention, Control | Non Intervention
Number analyzed (Participants) | 272 | 237
kg/m^2 | 16.4 (2.8) | 17.0 (2.4)
Statistical Analysis 1: Comparison: Educational Intervention, Control vs Non Intervention; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mixed-effects linear regression, adjusted for clustering within schools and children to assess the effect of intervention on changes in BMI over time

2. Secondary Outcome: Height
Time Frame: every two years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Educational Intervention, Control | Non Intervention
Number analyzed (Participants) | 272 | 237
m | 1.21 (0.06) | 1.19 (0.06)

3. Secondary Outcome: Father's Height
Time Frame: every two years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Educational Intervention, Control | Non Intervention
Number analyzed (Participants) | 272 | 237
m | 1.74 (0.07) | 1.75 (0.07)

4. Secondary Outcome: Mother's Height
Time Frame: every two years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Educational Intervention, Control | Non Intervention
Number analyzed (Participants) | 272 | 237
m | 1.61 (0.07) | 1.62 (0.07)

ADVERSE EVENTS:
Groups:
- Educational Intervention, Control: No untoward or unfavorable medical occurrence in a participants. There's no medication
Arm/Group | Educational Intervention, Control | Non Intervention
All-Cause Mortality (participants affected / at risk) | 0/237 | 0/272
Serious Adverse Events (participants affected / at risk) | 0/237 | 0/272
Other Adverse Events (participants affected / at risk) | 0/237 | 0/272

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No